CLINICAL TRIAL: NCT04228068
Title: A Home-Based Rehabilitation Program for Patients With Hip Fracture: A Pilot Randomized Trial
Brief Title: The Stronger at Home Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Mohammad Auais, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Mohammad Auais, PhD, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REH-721-18
Record Dates: First submitted 2020-01-03; First posted 2020-01-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The exercise program will be for the first 12 weeks after returning home. The intervention will be provided after patients return home. Each patient will receive 7 home visits in total over the intervention period by a physiotherapist (PT) and/or a physiotherapy assistant (PTA). Participants in the intervention group will receive a copy of the Toolkit before discharge from the hospital, and the study coordinator will walk them through it and explain what should be expected during the intervention period.
  Interventions: Other: Rehabilitation Program; Other: Pain self management
- Conventional care (Active Comparator): Usual care
  Interventions: Other: Conventional care

INTERVENTIONS:
Other: Rehabilitation Program — PT visits (two visits): The first visit will happen within a week of discharge. During this visit, the PT will assess participants, tailor the program to their needs, and coach them in carrying out the exercises at home. The last visit will be 12 weeks after the first. During this visit, the PT will reassess the participants and make adjustments to the program. The participants will be encouraged to continue exercising beyond the 12 weeks.
  The PTA will visit the participants' homes with the PT and will conduct additional solo visits every other week (i.e. 7 PTA visits in total, in 1st week and at 2, 4, 6, 8, 10, and 12 weeks). The PTA will facilitate and progress the exercise program as prescribed and directed by the PT and help in delivering the education component of the program.
  Arms: Intervention
Other: Pain self management — In addition to the exercise program, the intervention group will receive a pain self-management support tailored by the PT to the participants' needs.
  Arms: Intervention
Other: Conventional care — The control group will receive the usual care provided by the healthcare system.
  Arms: Conventional care

SUMMARY:
Hip fracture is a major health problem facing older adults. Hip fractures result in higher mortality, morbidity, and costs than all other osteoporotic fractures combined. When returning home following hip fracture surgery, patients are at high risk of adverse outcomes (e.g., secondary fractures, institutionalisation, and death).

Objectives: This study aims to finalize and pilot test a new program of care including a user-friendly toolkit containing a home-based physiotherapy exercise and pain management program to help community-dwelling older adults recover after hip fractures.

Methods: This study will be two stages: First, finalizing the program. The investigators have created a self-explanatory toolkit that includes an illustrated exercise program based on a critical analysis of previous programs for hip fracture patients. The investigators will organize focus groups and conduct semi-structured interviews with patients, caregivers, policymakers, and healthcare providers to review the program and provide feedback.

Second, conducting a feasibility study. The investigators will pilot the program in a randomized trial with community-dwelling hip fracture patients and compare the intervention with conventional care.

Expected Outcomes: While the number of hip fracture survivors is increasing, they are becoming frailer, and their functional recovery has not improved, making this study timely and relevant. With the current focus on helping older adults "age in place," the proposed project addresses a vital health system challenge: helping older hip fracture patients access proper rehabilitation, so they can stay independent in their homes.

ELIGIBILITY:
Inclusion Criteria:

* hip fracture patients who are 65 years or older
* being discharged to home or retirement home .

Exclusion Criteria:

* participants with a terminal illness or significant contraindications preventing exercising (e.g. rapidly progressing neurological disease),
* live away more than 30 km from the centre of the city, and
* cannot sign the consent form and no proxy available to sign.

Ages: 65 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the Lower Extremity Functional Scale (LEFS) | Change from baseline (before discharge) to 12 weeks post discharge to home (post intervention)
  The Lower Extremity Functional Scale is a patient-reported outcome measure that consists of 20 items. psychometric properties have been tested and established for different populations including patients after hip surgeries and lower extremity conditions. Score range is 0-80 with higher scores indicating better function.

SECONDARY OUTCOMES:
The Short Physical Performance Battery (SPPB) | Change from baseline (before discharge), to 12 weeks weeks post discharge to home
  The SPPB uses three tests to examine lower extremity physical performance: standing balance, gait speed, and chair-rising tests, and the total score is the sum of the three tests (0-12), with higher scores reflecting better physical function.

CONTACTS AND LOCATIONS:
Locations (1):
- Providence Care Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fairhall NJ, Dyer SM, Mak JC, Diong J, Kwok WS, Sherrington C. Interventions for improving mobility after hip fracture surgery in adults. Cochrane Database Syst Rev. 2022 Sep 7;9(9):CD001704. doi: 10.1002/14651858.CD001704.pub5. PMID 36070134